CLINICAL TRIAL: NCT06404879
Title: The Relationship Between Pre-operative Parental Anxiety Level and the Child's Anxiety Level and Its Effect on Postoperative Pain in Children Aged 2-6 Years Who Will Undergo Inguinal Area Surgery.
Brief Title: The Effect of Parental Anxiety Level on the Child's Anxiety Level and Postoperative Pain in Children Undergoing Surgery.
Status: Completed | Type: Observational
Sponsor: Giresun University (Other)
Responsible Party: Principal Investigator, Dilek Yeniay, Anesthesiology and Reanimation physician, Giresun University
Other Study IDs: 25.09.2023/07
Record Dates: First submitted 2024-04-29; First posted 2024-05-08 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Anxiety; Children
Keywords: children; anxiety; analgesia; pediatric; anaesthesia
MeSH Terms: conditions — Anxiety Disorders; Agnosia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- children group: Are between the ages of 2-6, are planned to undergo surgery under general anesthesia due to inguinal area pathology, No mental or neurological disorders in both mother and child No vision, hearing or speech problems in both mother and child Parents and children who volunteer to participate in the research will be included in the study.
  Those who did not volunteer to participate in the study, Undergoing surgery with a pathology other than the inguinal area, Having emergency surgery Children with pathologies (mental retardation, neurological problems, etc.) that may cause difficulty in communicating with both the family and the child will not be included in the study.
  Interventions: Other: determining scores with tests

INTERVENTIONS:
Other: determining scores with tests — Parents of children preparing for the operation will be given a child and family information form and STAI-I and STAI-II (State-Trait Anxiety Scale) scale forms and will be asked to fill them out themselves.
  An anesthesia technician blind to the content of the study will calculate and take notes on the children's anxiety levels, according to the m-YPAS (modified Yale Preoperative Anxiety) scale, in the preoperative waiting room (T1) and when the anesthesia ventilation mask is shown (T4).
  FLACC (Face, Legs, Activity, Cry, Consolabilityscale) scores and spO2, pulse values and complications such as nausea, vomiting and desaturation at the 5th, 10th, 20th and 30th minutes of all children taken to the recovery unit in the postoperative period will be recorded by the recovery unit nurse. . Children who are thought to have pain according to the FLACC score will be given 0.5 mg/kg meperidine as rescue analgesia and a note will be taken.

SUMMARY:
The aim of this prospective study is to investigate whether the anxiety levels of parents of children aged 2-6 years who will undergo inguinal area surgery have an effect on the child's preoperative anxiety level and postoperative pain level.

DETAILED DESCRIPTION:
Hospitalization of children for any health problem or treatment is a complex and difficult process that negatively affects the child and his family and creates stress. Surgical treatment in children can be planned or unplanned, minor or major, invasive or non-invasive, but every type of surgery is considered a stressful experience. Studies have shown that by controlling the anxiety and fear experienced in the preoperative period, children can achieve faster recovery in the postoperative period, better pain tolerance and earlier discharge. For this reason, we aim to contribute to the literature by investigating whether the anxiety levels of the parents of children aged 2-6 who will undergo inguinal area surgery affect the child's preoperative anxiety level and postoperative pain level.

ELIGIBILITY:
Inclusion Criteria:

* The child is between the ages of 2-6
* Patients scheduled for surgery under general anesthesia due to inguinal area pathology
* Surgery performed as planned
* There is no mental or neurological disorder in both the mother and the child.
* There are no vision, hearing or speech problems in both the mother and the child.
* Parents and children who volunteer to participate in the research
* Children with ASA I

Exclusion Criteria:

* Not volunteering to participate in the study (those for whom parental consent cannot be obtained)
* Those who underwent surgery with a pathology other than the inguinal area
* Having emergency surgery
* Children at risk with ASA 2 and above
* Having a pathology that may cause difficulty in communicating with both the family and the child (such as mental retardation, neurological problem).

Ages: 2 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Children who are planned to undergo surgery under general anesthesia due to inguinal area pathology
Sampling Method: Non-Probability Sample
Enrollment: 81 (Actual)
Dates: Start 2025-01-01 (Actual); Primary Completion 2025-04-01 (Actual); Study Completion 2025-05-16 (Actual)

PRIMARY OUTCOMES:
Anxiety level of parents | preoperative period
  It will be measured with STAI-I and STAI-II (State-Trait Anxiety Scale) scale forms.
Anxiety level of the child undergoing surgery | preoperative and intraoperative period
  According to the m-YPAS (modified Yale Preoperative Anxiety) scale, children's anxiety levels will be calculated in the preoperative waiting room (T1) and when the anesthesia ventilation mask is shown (T4).
Pain levels of children undergoing surgery | postoperative period
  Pain levels of all children taken to the recovery unit will be measured with the FLACC (Face, Legs, Activity, Cry, Consolabilityscale) score at the 5th, 10th, 20th and 30th minutes.

SECONDARY OUTCOMES:
heart rate | intraoperative period
  beats/min
heart rate | up to 8 hour postoperative
  beats/min
complication | up to 24 hour postoperative
  such as nausea, vomiting and desaturation

CONTACTS AND LOCATIONS:
Overall Officials: Dilek YENİAY, Principal Investigator — Department of Anesthesiolgy, Giresun University
Locations (1):
- Giresun Gynecology and Pediatrics Training Research Hospital, Giresun, Centre, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No